CLINICAL TRIAL: NCT05606172
Title: Adaptation of the Primary Care Intervention for PTSD for Children Aged 6 to 11
Brief Title: Adaptation of the PCIP for Children Aged 6 to 11
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We secured funding to run a cluster randomized trial and approval from the sponsor to transfer the money for this project to the new larger trial.
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Lauren Ng, PhD, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-001441
Record Dates: First submitted 2022-10-28; First posted 2022-11-04 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Post-Traumatic Stress Disorder in Children; Post-traumatic Stress Disorder
Keywords: Children; Primary Care; PTSD; Post Traumatic Stress Disorder; Randomized Pilot Feasibility Trial
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Mixed methods (qualitative and quantitative) randomized pilot feasibility trial (n=10 to treatment and 10 to waitlist control).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PCIP for youth aged 6 to 11 (Experimental): This arm will receive the adapted PCIP intervention lasting from 1-4 weeks, and will complete baseline, post treatment, 1-month, and 3-month follow up assessments.
  Interventions: Behavioral: Primary Care Intervention for PTSD (PCIP) Youth aged 6 -11
- Waitlist Treatment as Usual (Active Comparator): Receive standard care treatment and will complete baseline, post treatment, 1-month, and 3-month follow up assessments, and are offered PCIP treatment after conclusion of the study.
  Interventions: Behavioral: Waitlist Treatment as Usual

INTERVENTIONS:
Behavioral: Primary Care Intervention for PTSD (PCIP) Youth aged 6 -11 — This treatment ranges from 1-4 sessions which last 50 minutes per session. The first session will cover psychoeducation about PTSD symptoms in children that can be delivered to the parent or both the parent and child. The first session will also teach the parent and child a breathing technique to combat the physiological impact of PTSD in children. The subsequent sessions will be tailored to meet the needs of the child's most distressing PTSD symptom cluster including hyper arousal, negative changes in cognition and mood, avoidance, re-experiencing. Each session contains coping skills that the parent and child can learn together. There is also material for parents to address behavior problems in youth. This treatment will be delivered via telehealth.
  Arms: PCIP for youth aged 6 to 11
Behavioral: Waitlist Treatment as Usual — Will receive treatment as usual at local clinic and are provided information on free or low cost mental health care referrals in the Los Angeles Area.
  Arms: Waitlist Treatment as Usual

SUMMARY:
This study will implement a brief Post-traumatic Stress Disorder (PTSD) intervention for children, the Primary Care Intervention for PTSD (PCIP) delivered through telehealth (computer or smartphone delivery), to 10 youth age 6-11 and their caregivers.

Mixed methods (qualitative and quantitative) randomized pilot feasibility trial (n=10 to treatment and 10 to waitlist control) to refine the intervention, study procedures, and explore effectiveness.

Following RE-AIM guidelines, the investigators will assess:

1. Reach: patient participation in intervention delivery (out of all those asked to participate) and retention rate (out of all those who consented to participate and completed at least two intervention sessions)
2. Adoption: patients and their parents/guardians will complete screening and intervention satisfaction ratings.

To understand patient experiences with the intervention and to identify and explain positive or negative treatment mechanisms or effects, the investigators will conduct post-intervention semi-structured interviews with the participating patients, their parents/guardians, and with providers.

This treatment ranges from 1-4 sessions which last 50 minutes per session. The first session will cover psychoeducation about PTSD symptoms in children that can be delivered to the parent or both the parent and child. The first session will also teach the parent and child a breathing technique to combat the physiological impact of PTSD in children. The subsequent sessions will be tailored to meet the needs of the child's most distressing PTSD symptom cluster including hyper arousal, negative changes in cognition and mood, avoidance, re-experiencing. Each session contains coping skills that the parent and child can learn together. There is also material for parents to address behavior problems in youth. This treatment will be delivered via telehealth.

ELIGIBILITY:
Inclusion Criteria:

1. Patient referred to the SHARK Program
2. Patients must be at least 6 years old
3. The patient's legal guardian is able and willing to provide informed consent for the patient to participate in the study;
4. Patient is able to complete study activities in English.

Exclusion Criteria:

1. Suicidal ideation with a plan within the last two weeks or a suicide attempt within the past 30 days;
2. Inability to provide informed consent or assent, and/or complete procedures in English.
3. Patient is over the age of 11

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Change in PTSD Knowledge | Day 0 baseline, 3 months
  Changes in levels of PTSD Knowledge measured by the PTSD Knowledge Test (0-14, higher scores indicating more PTSD knowledge)
Change in Self-Reported Arousal | Day 0 baseline, 3 months
  Changes in PTSD related arousal levels measured by the Self-Assessment Manikin (SAM; 0-24, higher scores indicating higher arousal)
Intervention Acceptability | 1 month
  Qualitative interviews will include questions regarding acceptability of treatment including treatment via telehealth and barriers to treatment.
Intervention Engagement | 1 month
  Data will be collected regarding participant completion of therapy, no show rates, and attendance.
Intervention Implementation | 1 month
  Study therapists will complete qualitative interviews regarding intervention delivery feasibility and study protocols.

SECONDARY OUTCOMES:
Change in PTSD and Trauma Symptoms | Day 0 baseline, 3 months
  Changes in trauma related symptoms measured by Child and Adolescent Trauma Screen (CATS) Self Report and Caregiver report (total 0-60, Higher scores indicated greater symptom severity).
Change in Depression Symptoms | Day 0 baseline, 3 months
  Changes in depression symptoms measured by the Center for Epidemiologic Studies Depression Scale (CES-DC) Self Report (total 0-60, Higher scores indicate higher symptom severity).
Change in Anxiety Symptoms | Day 0 baseline, 3 months
  Changes in anxiety symptoms measured by the Revised Children's Anxiety and Depression Scale (RCADS) Self Report (total 0-141, Higher scores indicating higher symptom severity).
Change in Positive Parenting Practices | Day 0 baseline, 3 months
  Changes in positive Parenting Practices measured by the Alabama Parenting Questionnaire (total 45-210, Higher scores indicating higher instances more positive parenting).

CONTACTS AND LOCATIONS:
Overall Officials: Lauren C Ng, PhD, Principal Investigator — UCLA Psychology
Locations (1):
- University of California Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No